CLINICAL TRIAL: NCT03747211
Title: The ATOM Study: Asthma Severity in Women: The Influence of Training and Menopause
Brief Title: Asthma Severity in Women: The Influence of Training and Menopause
Acronym: ATOM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues recruiting participants during COVID-19
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Backer, Professor, Dr.med, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATOM
Record Dates: First submitted 2018-11-09; First posted 2018-11-20 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Late-Onset Asthma
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, outcome assessor blinded, controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Concealed computer generated allocation via REDCap
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise intervention (Experimental): Aerobic exercise by high intensity interval training, 3 times per week for 12 weeks
  Interventions: Behavioral: Aerobic exercise
- Control group (No Intervention): No intervention for 12 weeks

INTERVENTIONS:
Behavioral: Aerobic exercise — High Intensity Interval Training (HIIT)
  Arms: Aerobic exercise intervention

SUMMARY:
Introduction: Late-onset asthma in women is characterized by poor disease control and reduced quality of life despite intensive treatment with inhaled steroid and beta2-agonist. The condition is further worsened at menopause due to the loss of estrogen leading to increased asthma exacerbation frequency, increased airway inflammation and decreased lung function. Exercise training may increase disease control of asthma patients, but to what extent the same effect is seen in postmenopausal women with late-onset asthma is unknown. These asthma patients represent a phenotype that is characterized by low eosinophilic airway inflammation, severe symptoms, moderate obesity and poor response to conventional medicine. Thus, our hypothesis is that regular physical exercise is especially associated with an improvement in asthma control in this phenotype. The aim of this project is to test this hypothesis and to assess whether an improvement is associated with reduced local and systemic inflammation, change in heart function, lung function and/or body composition.

Study design: 40 postmenopausal women with late-onset asthma are recruited via the outpatient clinic at the Respiratory Department at Bispebjerg Hospital and through advertisement. The participants are randomized 1:1 into two groups. One group performs supervised exercise training (spinning) three times per week for 12 weeks while the other group is a control group. Before and after the intervention asthma control, local and systemic inflammation, heart function and body composition is measured.

Results: Analysis will be performed to detect changes within and between the groups before and after intervention. Primary outcome is change in ACQ (Asthma Control Questionnaire). Local and systemic inflammation is measured by changes in bronchial challenge to methacholine, sputum cell count and blood tests. Furthermore, secondary outcomes include change in heart function measured by stress-echocardiography and change in body composition measured by Dual-energy X-ray absorptiometry (DEXA).

Conclusion: There are to date no prospective studies that can support recommendations containing asthma rehabilitation with supervised regular physical activity for postmenopausal women. Thus, this study will provide novel understanding of the importance of physical activity in a chronic disease such as asthma.

DETAILED DESCRIPTION:
Overall study design

The study is a single-blinded randomized controlled intervention study. Forty postmenopausal women with late-onset asthma (>16 years at debut) are recruited from the asthma outpatient-clinic at Bispebjerg Hospital or other hospital/practitioner in the region and/or by advertisement. The participants are block-randomized into two groups of 20, where one group is control and the other undergoes a period of regular exercise training. The investigators will be blinded and will not know whether the subjects have trained or not.

Detailed study design

Participants allocated to the exercise training group undergo a training intervention consisting of 45 minutes of intermittent high intensity aerobic spinning training three times per week for 12 weeks. Participants allocated to the control group will continue usual care without training. No changes to current treatment will be made by the investigators on any of the groups.

The training will consist of short periods of high intensity intervals where subjects reach above 80% of maximal oxygen consumption. Spinning sessions will be fully supervised by trained instructors with a bachelor of sports and science or bachelor of medicine and conducted in the Department of Nutrition, Exercise and Sports, University of Copenhagen. Subjects will wear heart rate monitors to ensure adherence to the training protocol. Within two weeks, before and after the intervention, participants from both groups undergo 3 days of testing.

To ensure equal compliance with asthma medication both groups will receive daily electronic reminders. Once a week, all participants will be asked about their compliance to their medication.

ELIGIBILITY:
Inclusion Criteria:

* Late onset asthma (Debut ≥ 16 years of age)
* ACQ ≥ 1.25
* Daily treatment for asthma (GINA 2 and above)
* Age 45 - 75
* Postmenopausal defined as no menstruation for 6 months, Serum Follicle stimulating hormone >20 International Units per Liter and P-Estradiol nmol/L <0.09
* BMI 25 - 35
* Positive bronchial challenge to methacholine, mannitol or positive reversibility to beta2-agonist now or historically
* Untrained (no participation in vigorous exercise for more than 1 hour per week during the last 2 months)
* Capable of exercising on a bike

Exclusion Criteria:

* Unable to speak and understand Danish or English.
* Current or former smokers (>6 months cessation) with >20 years of daily smoking with 20 cigarettes per day.
* Other respiratory disease of clinical significance
* Cardiovascular: Unstable ischemic heart disease, myocardial infarction within the last 12 months, symptomatic heart failure (EF <40%), symptomatic heart arrhythmia (documented with ECG), uncontrolled hypertension (>155/100)
* Any disorder that is not stable and in the opinion of the investigator could affect the safety of the subject throughout the study
* Subjects, who by investigators determination, will not be able to adhere to study protocol

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Asthma control - Asthma Control Questionnaire (ACQ) | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in Asthma Control Questionnaire (ACQ) 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use)

SECONDARY OUTCOMES:
Heart Rate Variability | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in:
  - Heart rate variability
Heart rhytm | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in:
  - Heart rhythm
Heart Rate | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in:
  - electrocardiography
Heart function - Strain | -21 to 0 days before intervention and 0 to 14 days post intervention
  Measured by stress-echocardiography
  - Strain
Heart function - Ejection fraction | -21 to 0 days before intervention and 0 to 14 days post intervention
  Measured by stress-echocardiography
  - Ejection fraction
Heart function - Tricuspid annular plane systolic excursion | -21 to 0 days before intervention and 0 to 14 days post intervention
  Measured by stress-echocardiography
  - Tricuspid annular plane systolic excursion
Heart function - Right ventricular function | -21 to 0 days before intervention and 0 to 14 days post intervention
  Measured by stress-echocardiography
  - Right ventricular function
Heart function - Pulmonary pressure | -21 to 0 days before intervention and 0 to 14 days post intervention
  Measured by stress-echocardiography
  - Pulmonary pressure
Heart function - Lung covered cor | -21 to 0 days before intervention and 0 to 14 days post intervention
  Measured by stress-echocardiography
  - Lung covered cor
Heart function - Blood pressure | -21 to 0 days before intervention and 0 to 14 days post intervention
  Blood pressure
Heart function - Cardiac output | -21 to 0 days before intervention and 0 to 14 days post intervention
  Cardiac output
Heart function - Stroke volume | -21 to 0 days before intervention and 0 to 14 days post intervention
  Stroke volume
Heart function - Total peripheral resistance | -21 to 0 days before intervention and 0 to 14 days post intervention
  Total peripheral resistance
Systemic inflammation - Leukocytes + differential cell count count | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Leukocytes + differential cell count count
Systemic inflammation - Interleukin 6 | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Interleukin 6
Systemic inflammation - Interleukin 8 | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Interleukin 8
Systemic inflammation | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Other interleukins
Systemic inflammation - Tumor Necrosis Factor alpha | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Tumor Necrosis Factor alpha
Systemic inflammation - Total immunoglobulin E, Specific immunoglobulin E | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  * Total immunoglobulin E
  * Specific immunoglobulin E
Systemic inflammation - high sensitivity c reactive protein | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - high sensitivity c reactive protein
Local airway inflammation - Sputum cell count | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Sputum cell count
Local airway inflammation - Fraction of exhaled nitric oxide | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Fraction of exhaled nitric oxide
Local airway inflammation - Hyperreactivity to inhaled methacholine | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Hyperreactivity to inhaled methacholine
Body Composition | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Total body fat
Body Composition | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Lean body mass
Body Composition | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Muscle mass
Body Composition | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Weight
Microbiome | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in the microbiota in sputum, oral cavity and nasal cavity before and after the training intervention
Compliance - Foster score | -21 to 0 days before intervention and 0 to 14 days post intervention
  Change in
  - Foster score Answers describe last weeks medicine use. Answers range form 0/7 - 7/7 with low values being worse.
Other asthma related questionnaires - Nijmegen questionnaire | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Nijmegen questionnaire Values range from 0-64 and values below 20 are considered normal.
Other asthma related questionnaires - Mini Asthma Quality of Life Questionnaire (miniAQLQ) | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Mini Asthma Quality of Life Questionnaire (miniAQLQ) 7-point Likert scale (7 = not impaired at all - 1 = severely impaired).
Other asthma related questionnaires - Hospital Anxiety and Depression Scale (HADS) 2 items with 7 questions regarding anxiety and depression. (0 = no sign of depression/anxiety, 21 = maximal signs of anxiety/depression) | -21 to 0 days before intervention and 0 to 14 days post intervention
  Changes in
  - Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, Physician, Principal Investigator — Respiratory Research Unit, Bispebjerg Hospital
Locations (1):
- Respiratory research unit, Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data that support the results of this study will be made available immediately, with no end date, after deidentification and upon reasonable request.
Time Frame: Immediately after publication with no end date.
Access Criteria: Data will be made available upon reasonable request to achieve the aims of the reasonable request.

REFERENCES:
- [Derived] Hansen ESH, Rasmusen HK, Hostrup M, Hellsten Y, Backer V. The effect of aerobic exercise training on asthma control in postmenopausal women (ATOM): a randomized controlled pilot study. Eur Clin Respir J. 2023 Sep 4;10(1):2251256. doi: 10.1080/20018525.2023.2251256. eCollection 2023. PMID 37674777
- [Derived] Hansen ESH, Hostrup M, Rasmusen HK, Hellsten Y, Backer V. Effect of aerobic exercise training on asthma control in postmenopausal women (the ATOM-study): protocol for an outcome assessor, randomised controlled trial. BMJ Open. 2021 Apr 22;11(4):e049477. doi: 10.1136/bmjopen-2021-049477. PMID 33888532